CLINICAL TRIAL: NCT02449902
Title: A Phase 1, Randomized, Double-blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of TX-12-004-HR in Postmenopausal Women With Symptoms of Vulvar and Vaginal Atrophy (VVA)
Brief Title: TXV13-01 Estradiol Vaginal Softgel Capsules in Treating Postmenopausal Women With Symptoms of Vulvar and Vaginal Atrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TherapeuticsMD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TXV13-01
Record Dates: First submitted 2015-05-18; First posted 2015-05-20 (Estimated); Results first posted 2015-12-14 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-11

CONDITIONS: Menopause; Vulvovaginal Atrophy; Painful Intercourse; Dyspareunia
Keywords: VVA; Postmenopausal; Painful Sex
MeSH Terms: conditions — Dyspareunia | interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment 1 (Active Comparator): Estradiol 10 μg vaginal softgel capsule
  Interventions: Drug: Estradiol
- Treatment 2 (Placebo Comparator): Placebo vaginal softgel capsule
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Estradiol — 1 10 µg capsule inserted vaginally for 14 days.
  Other Names: 17β-estradiol
  Arms: Treatment 1
Drug: placebo — 1 placebo capsule inserted vaginally for 14 days.
  Arms: Treatment 2

SUMMARY:
The study was designed to evaluate the efficacy and safety of TX-12-004-HR 10 μg in treating moderate to severe symptoms of vaginal atrophy associated with menopause after 14 days of treatment, and to estimate the effect size and variability of vulvovaginal atrophy endpoints. In addition, the systemic exposure to estradiol from single and multiple doses of TX-12-004-HR was to be investigated.

DETAILED DESCRIPTION:
This study was a randomized, double-blind, placebo-controlled trial to evaluate safety and efficacy of the TX-12-004-HR formulation in reducing moderate to severe symptoms of vaginal atrophy associated with menopause and to investigate the systemic exposure to estradiol following once daily intravaginal administrations of TX-12-004-HR for 14 days.

Postmenopausal subjects who met the study entry criteria were randomized to one of two treatment groups (TX-12-004-HR or Placebo). During the Screening period subjects were asked to self-assess the symptoms of vulvar and/or vaginal atrophy, including vaginal dryness, vaginal and/or vulvar irritation/itching, dysuria, vaginal pain associated with sexual activity and vaginal bleeding associated with sexual activity. Subjects with at least one self-assessed moderate to severe symptom of vulvar and/or vaginal atrophy identified by the subject as being most bothersome to her were eligible to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Be a female between 40 and 75 years (at the time of randomization) who is willing to participate in the study, as documented by signing the informed consent form.
2. Be a postmenopausal woman. Postmenopausal is defined with at least 12 months of spontaneous amenorrhea or 12 months post bilateral oophorectomy, with or without hysterectomy (documented by an operative report or patient reported). Women ≥ 60 years of age who have had a hysterectomy without bilateral oophorectomy prior to natural menopause are considered menopausal.
3. Have a baseline evaluation requirements:

   * ≤5% superficial cells on vaginal smear cytology
   * Vaginal pH > 5.0
   * Estradiol level ≤ 50 pg/ml
   * At least one self-assessed moderate to severe symptom of vulvar and/or vaginal atrophy from the following list that is identified by the subject as being most bothersome to her:

     * Vaginal dryness
     * Vaginal pain associated with sexual activity
     * Vaginal and/or vulvar irritation/itching
     * Dysuria
     * Vaginal bleeding associated with sexual activity (absence vs. presence)
4. Have a Body Mass Index (BMI) less than or equal to 34 kg/m2. (BMI values should be rounded to the nearest integer [e.g., 34.4 rounds down to 34, while 26.5 rounds up to 27]).
5. Be willing to abstain from using products (other than study medication) that contain estrogen throughout study participation.
6. Be judged by the Principal Investigator or Sub-investigator as being in otherwise generally good health based on a pre-study medical evaluation performed within 28 days prior to the initial dose of study medication. The medical evaluation findings must include:

   * a normal or non-clinically significant physical examination, including vital signs (sitting blood pressure, heart rate, respiratory rate and temperature).
   * a normal or non-clinically significant pelvic examination.
   * a mammogram that shows no sign of significant disease (can be performed within previous 9 months prior to initial dose of study medication). An acceptable mammogram is defined as a mammogram in which no masses or other findings are identified that is suspicious of malignancy. The site must obtain a copy of the official report for the subject's study file, and it must be verified that the mammogram itself is available if needed for additional assessment.
   * a normal or non-clinically significant clinical breast examination. An acceptable breast examination is defined as no masses or other findings identified that are suspicious of malignancy.
   * a normal Screening Papanicolaou ("Pap") smear (ASCUS with high risk- human papillomavirus (HPV) negative is acceptable).
   * within normal limits or non-clinically significant laboratory evaluation results
   * sitting systolic blood pressure ≤140 mmHg and diastolic blood pressure ≤90 mmHg at Screening. A subject may be taking up to two antihypertensive medications.
7. Be willing to abstain from sexual activity and use of vaginal douching within 24 hours prior to screening and Visit 3 vaginal pH measurements.

Exclusion Criteria:

1. Be currently hospitalized.
2. Have a history of thrombosis of deep veins or arteries or a thromboembolic disorder.
3. Have a history of coronary artery or cerebrovascular disease.
4. Have a history of liver or kidney dysfunction/disorder.
5. Have a history of gallbladder dysfunction/disorders (e.g., cholangitis, cholecystitis), unless gallbladder has been removed.
6. Have a history of diabetes, thyroid disease (subjects with diet-controlled diabetes, or controlled hypothyroid disease at Screening are not excluded), or any other endocrinological disease.
7. Have a history of estrogen-dependent neoplasia.
8. Have a history of atypical ductal hyperplasia of the breast.
9. Have a history of undiagnosed vaginal bleeding.
10. Have a vaginal infection requiring treatment
11. Have any history of endometrial hyperplasia or uterine/endometrial, breast or ovarian cancer.
12. Have any history of other malignancy within the last 5 years, with the exception of basal cell (excluded if within 1 year) or non-invasive squamous cell (excluded if within 1 year) carcinoma of the skin.
13. Have a history of any other cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, psychological, or musculoskeletal disease or disorder that is clinically significant in the opinion of the Principal Investigator or Medical Sub-Investigator.
14. Have contraindication to estrogen therapy or allergy to the use of estradiol or any components of the investigational drugs.
15. Use 15 or more cigarettes per day.
16. Have a history of drug and/or alcohol abuse within one year of start of study.
17. Have used, within 28 days prior to Screening, or plan to use during the study, any prescription or over-the-counter (OTC) medications (including herbal products) that would be expected to interact with estradiol therapy.
18. Use of any type of vaginal preparation (including lubricants and moisturizers) within 14 days prior to Screening.
19. Have used estrogen alone or estrogen/progestin for any of the following time periods:

    * Vaginal hormonal products (rings, creams, gels) within 3 months prior to Screening.
    * Transdermal estrogen alone or estrogen/progestin products within 8 weeks prior to Screening.
    * Oral estrogen and/or progestin therapy within 8 weeks prior to Screening.
    * Progestational implants, estrogen or estrogen/progestational injectable drug therapy within 3 months prior to Screening.
    * Estrogen pellet therapy or progestational injectable drug therapy within 6 months prior to Screening.
    * Percutaneous estrogen lotions/gels within 8 weeks prior to Screening.
    * Oral, topical, vaginal, patch, implantable or injectable androgen therapy within 8 weeks prior to Screening.
20. Have any reason which, in the opinion of the Principal Investigator or Medical Sub-Investigator, would prevent the subject from safely participating in the study or complying with protocol requirements.
21. Have contraindication to any planned study procedure (e.g., blood collection).
22. Have participated in another clinical trial within 30 days prior to screening, have received an investigational drug within the three months prior to the initial dose of study medication, or be likely to participate in a clinical trial or receive another investigational medication during the study.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shelli Graham, PhD, Study Director — TherapeuticsMD
Locations (1):
- Avail Clinical Research, DeLand, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- TX-12-004-HR 10μg: Active treatment group. Subjects self-administered the active treatment, a single capsule of 10 μg Estradiol, intravaginally once daily for 14 days.
- Placebo: Control treatment group. Subjects self-administered the control treatment, a single placebo matching capsule, intravaginally once daily for 14 days.
Period: Overall Study
Arm/Group | TX-12-004-HR 10μg | Placebo
Started | 24 | 26
Completed | 24 | 24
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Estradiol 10 μg Daily for 14 Days: Active treatment group. Subjects self-administered the active treatment, a single capsule of 10 μg Estradiol, intravaginally once daily for 14 days.
- Placebo Daily for 14 Days: Control treatment group. Subjects self-administered the control treatment, a single placebo matching capsule, intravaginally once daily for 14 days.
- Total: Total of all reporting groups
Arm/Group | Estradiol 10 μg Daily for 14 Days | Placebo Daily for 14 Days | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (5.7) | 62.3 (7.0) | 62.3 (6.4)
Sex/Gender, Customized [Number; unit: participants]
  Female | 24 | 26 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 21 | 24 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 26 | 50
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 26.4 (3.9) | 27.2 (3.3) | 26.8 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: Analysis of Change From Baseline to Day 15 in Maturation Index of the Vaginal Cell Type (Parabasal Cells)
Time Frame: Baseline to 15 days post-treatment
Measure: Least Squares Mean (Standard Error); unit: Percentage of Parabasal Cells
Groups:
- TX-12-004-HR 10μg: Active treatment group.
- Placebo: Control treatment group.
Arm/Group | TX-12-004-HR 10μg | Placebo
Number analyzed (Participants) | 24 | 24
Percentage of Parabasal Cells | -54.4 (4.6) | -4.8 (4.6)
Statistical Analysis 1: Comparison: TX-12-004-HR 10μg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA

2. Primary Outcome: Analysis of Change From Baseline to Day 15 in Maturation Index of the Vaginal Cell Type (Superficial Cells)
Time Frame: Baseline to 15 days post-treatment
Measure: Least Squares Mean (Standard Error); unit: Percentage of Superficial Cells
Arm/Group | TX-12-004-HR 10μg | Placebo
Number analyzed (Participants) | 24 | 24
Percentage of Superficial Cells | 35.2 (4.7) | 8.8 (4.7)
Statistical Analysis 1: Comparison: TX-12-004-HR 10μg vs Placebo; Test type: Superiority or Other; p = 0.0002, ANOVA

3. Primary Outcome: Analysis of Change From Baseline to Day 15 in Maturation Index of the Vaginal Cell Type (Intermediate Cells)
Time Frame: Baseline to 15 days post-treatment
Measure: Least Squares Mean (Standard Error); unit: Percentage of Intermediate Cells
Arm/Group | TX-12-004-HR 10μg | Placebo
Number analyzed (Participants) | 24 | 24
Percentage of Intermediate Cells | 18.7 (4.7) | -3.5 (4.7)
Statistical Analysis 1: Comparison: TX-12-004-HR 10μg vs Placebo; Test type: Superiority or Other; p = 0.0017, ANCOVA

4. Primary Outcome: Analysis of Change From Baseline to Day 15 in Vaginal pH
Time Frame: Baseline to 15 days post-treatment
Measure: Least Squares Mean (Standard Error); unit: pH
Arm/Group | TX-12-004-HR 10μg | Placebo
Number analyzed (Participants) | 24 | 24
pH | -0.97 (0.1) | -0.34 (0.1)
Statistical Analysis 1: Comparison: TX-12-004-HR 10μg vs Placebo; Test type: Superiority or Other; p = 0.0002, ANCOVA

5. Primary Outcome: Analysis of Change From Baseline to Day 15 in Severity of the Most Bothersome Vulvar and Vaginal Atrophy (VVA) Symptom
Description: The severity of the most bothersome VVA symptom was self-assessed by each subject using a VVA questionnaire. The questionnaire has a 4-point scoring scale with: None=0, Mild=1, Moderate=2, and Severe=3. The lower the score, the least bothersome it is to the subject.
Time Frame: Baseline to 15 days post-treatment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TX-12-004-HR 10μg | Placebo
Number analyzed (Participants) | 24 | 24
units on a scale | -1.043 (0.2) | -1.042 (0.2)
Statistical Analysis 1: Comparison: TX-12-004-HR 10μg vs Placebo; Test type: Superiority or Other; p = 0.9951, ANOVA

6. Primary Outcome: Analysis of Change From Baseline to Day 15 in Vaginal Bleeding Associated With Sexual Activity
Description: Total number (N=10) of participants analyzed within each treatment group who were sexually active at both Baseline and Day 15 and provided a response at both visits.
Time Frame: Baseline to 15 days post-treatment
Population: Total number (N=10) of participants analyzed within each treatment group who were sexually active at both Baseline and Day 15 and provided a response at both visits.
Measure: Number; unit: participants
Arm/Group | TX-12-004-HR 10μg | Placebo
Number analyzed (Participants) | 10 | 10
participants
  Bleeding/ No Bleeding (Success) | 2 | 1
  Bleeding/ Bleeding (Failure) | 0 | 3
  No Bleeding/ Bleeding (Failure) | 0 | 1
  No Bleeding/ No Bleeding (No Change) | 8 | 5
Statistical Analysis 1: Comparison: TX-12-004-HR 10μg vs Placebo; Test type: Superiority or Other; p = 0.1429, Fisher Exact

7. Primary Outcome: Analysis of Change From Baseline to Day 15 in Investigator Assessment of the Vaginal Mucosa (Assessment of Vaginal Color)
Description: Outcome was measured by using a severity scale. No Atrophy is pink in color (0). Mild atrophy is lighter in color (1). Moderate atrophy is pale in color (2). Severe atrophy is transparent, either no color or inflamed (3).
Time Frame: Baseline to 15 days post-treatment
Population: All participants receiving at least one day of study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TX-12-004-HR 10μg | Placebo
Number analyzed (Participants) | 24 | 24
units on a scale | -0.199 (0.1) | -0.009 (0.1)
Statistical Analysis 1: Comparison: TX-12-004-HR 10μg vs Placebo; Test type: Superiority or Other; p = 0.1945, ANCOVA

8. Primary Outcome: Analysis of Change From Baseline to Day 15 in Investigator Assessment of the Vaginal Mucosa (Assessment of Vaginal Epithelial Integrity)
Description: Outcome was measured by using a severity scale. No Atrophy=normal(0). Mild atrophy=vaginal surface bleeds with scraping(1). Moderate atrophy=vaginal surface bleeds with light contact(2). Severe atrophy=vaginal surface has petechiae before contact and bleeds with light contact(3).
Time Frame: Baseline to 15 days post-treatment
Population: All participants receiving at least one day of study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TX-12-004-HR 10μg | Placebo
Number analyzed (Participants) | 24 | 24
units on a scale | -0.342 (0.1) | 0.176 (0.1)
Statistical Analysis 1: Comparison: TX-12-004-HR 10μg vs Placebo; Test type: Superiority or Other; p = 0.0001, ANCOVA

9. Primary Outcome: Change From Baseline to Day 15 in Investigator Assessment of the Vaginal Mucosa (Assessment of Vaginal Epithelial Surface Thickness)
Description: Outcome was measured by using a severity scale. No Atrophy has rogation and elasticity of vault(0). Mild atrophy has poor rogation with some elasticity noted of vaginal vault(1). Moderate atrophy is smooth, some elasticity of vaginal vault(2). Severe atrophy is smooth, no elasticity, constriction of the upper one third of vagina or loss of vaginal tone (cystocele and rectocele)(3).
Time Frame: Baseline to 15 days post-treatment
Population: All participants receiving at least one day of study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 24 | 24
units on a scale | -0.034 (0.1) | -0.133 (0.1)
Statistical Analysis 1: Comparison: Treatment 1 vs Treatment 2; Test type: Superiority or Other; p = 0.1820, ANCOVA

10. Primary Outcome: Analysis of Change From Baseline to Day 15 in Investigator Assessment of the Vaginal Mucosa (Assessment of Vaginal Secretions)
Description: Outcome was measured by using a severity scale. No Atrophy has normal clear secretions noted on vaginal walls(0). Mild atrophy has superficial coating of secretions, difficulty with speculum insertion(1). Moderate atrophy is scant not covering the entire vaginal vault, may need lubrication with speculum insertion to prevent pain(2). Severe atrophy has none, inflamed, ulceration noted, need lubrication with speculum insertion to prevent pain(3).
Time Frame: Baseline to 15 days post-treatment
Population: All participants receiving at least one day of study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TX-12-004-HR 10μg | Placebo
Number analyzed (Participants) | 24 | 24
units on a scale | -0.643 (0.1) | -0.274 (0.1)
Statistical Analysis 1: Comparison: TX-12-004-HR 10μg vs Placebo; Test type: Superiority or Other; p = 0.0401, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 14 days (study duration). Subjects with AEs that were ongoing at study completion or study withdrawal were followed until resolution or for 30 days after the last dose of study medication.
Description: Investigators evaluated adverse events for duration, severity, seriousness, causal relationship to the investigational drug and reviewed laboratory assessments per protocol.
Groups:
- TX-12-004-HR: Active treatment group.
Arm/Group | TX-12-004-HR | Placebo
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 13/24 | 4/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TX-12-004-HR (N=24) | Placebo (N=26)
Blood pressure increased (Blood and lymphatic system disorders) | 1 | 0
Eye Contusion (Eye disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Vaginal dysplasia (Reproductive system and breast disorders) | 4 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 2
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 1 | 0
Hot flush (Reproductive system and breast disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators may publish their own data provided that the information is reviewed by the Sponsor. Otherwise, publication of the outcome and results of the study will be the sole domain of Sponsor, and publication of the study results by the Institution or Principal Investigator is not permitted, except with the Sponsor's prior written consent.